CLINICAL TRIAL: NCT01493232
Title: Comparing Patient Satisfaction & Stress Distribution on Mandibular Ridge by Three Posterior Occlusal Scheme in Complete Denture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Javad Shirani, Mohammad Javad Shirani, Isfahan University of Medical Sciences, Faculty of dentistry,Dnt.mui.ac.ir, Perincipal investigator, Dental student., Isfahan University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 190052; IRCT201110097749N1 (Other Grant/Funding Number: Medical Uuniversity of Isfehan 1244003)
Record Dates: First submitted 2011-12-12; First posted 2011-12-15 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Edentulous
Keywords: Lingualized occlusion; Complete denture occlusion; Fully bilateral balanced occlusion; Patient satisfaction of complete denture
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Denture, edentulous patient, treatment (Experimental): Dentures with different type of occlusion
  Interventions: Other: buccalized occlusion
- Denture, Edentulous patient, treatment (Experimental): Dentures with different type of occlusion
  Interventions: Other: buccalized occlusion

INTERVENTIONS:
Other: buccalized occlusion — Making a set of complete denture with new Buccalized Occlusion that is different from current occlusion in my country. In this type just buccal casps of mandibular teeth will be connect to the central fossa of maxillary teeth and lingual casps have not contact.
  Other Names: K06.9; Disorder of gingiva and edentulous alveolar ridge, unspecified

SUMMARY:
In this randomized clinical trial to compare the patients' satisfaction of complete dentures with different occlusal forms, after simple randomized sampling of 15 participant that will be signed informed consent and their latest teeth was extracted 3 month ago, will be selected. For each participant, it will be made 3 set of complete dentures that are variable in occlusion only. During the study, dissatisfied participants can leave it. Each set will be inserted for 1month in 5 participant randomly. The participants will be examined in two stages, after a day and after a week. At the end of month the questionaire will be filled out and the pressure under the mandibular denture base will be measured with the pressure sensors. Then the second and third denture will be inserted simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* edentulous patients
* at least 3 month ago the latest teeth was extracted
* ideal jaw relation
* signing the informed consent

Exclusion Criteria:

* uncontrolled systemic disease
* mentally problem
* dissatisfaction for keeping on the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-03 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Patients' Satisfaction | 1 year
  method of measurement is Questionair

SECONDARY OUTCOMES:
Patients' Dissatisfaction | 1 year
  method of measurement Examination and Questionair

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Mosharraf, Prosthodontics Specialist, Study Chair — Medical University of Isfahan
Locations (1):
- Department of Prosthodontics, Faculty of Dentistry, Medical University of Isfahan, Isfahan, Isfahan, Iran

REFERENCES:
- [Derived] Shirani M, Mosharraf R, Shirany M. Comparisons of patient satisfaction levels with complete dentures of different occlusions: a randomized clinical trial. J Prosthodont. 2014 Jun;23(4):259-66. doi: 10.1111/jopr.12101. Epub 2013 Oct 19. PMID 24138344
- See also: Department of Research and Technology, Medical University of Isfahan, Iran — http://researches.mui.ac.ir